CLINICAL TRIAL: NCT04140630
Title: Exposure to Second-hand Aerosols Emitted by Use of Electronic Cigarettes in Real-life Conditions
Brief Title: Exposure to E-cigarette Aerosols in Real-life Conditions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Català d'Oncologia (Other)
Collaborators: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); University of Stirling (Other); Hellenic Cancer Society (Other); Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Other Study IDs: TackSHS WP8 Observational
Record Dates: First submitted 2019-10-01; First posted 2019-10-28 (Actual); Last update posted 2019-10-28 (Actual); Status verified 2019-10

CONDITIONS: Passive Exposure to Electronic Cigarette Aerosols
Keywords: vaping; electronic cigarette; passive exposure
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- E-cigarette users and bystanders: Households with one e-cigarette user (adult (18 years old and above); e-cigarette exclusive user for at least 1 month; daily use of e-cigarettes inside home; cohabiting with at least one non-tobacco product nor e-cigarette user; other household members should not be users of any tobacco products or e-cigarettes) and one bystander cohabiting with the user
  Interventions: Other: No intervention
- Conventional cigarette smokers and bystanders: Households with one smoker (adult (18 years old and above; manufactured cigarette exclusive smoker for at least 6 months; daily smoking inside home; cohabiting with at least one non-tobacco product nor e-cigarette user; other household members should not be users of tobacco products or e-cigarettes) and one bystander cohabiting with the smoker
  Interventions: Other: No intervention
- Heated tobacco product users and bystanders: Households with one user of the heated tobacco product, HTP (adult (18 years old and above; • HTP exclusive user for at least 1 month; daily use of HTP inside home; cohabiting with at least one non-tobacco product nor e-cigarette user; other household members should not be users of tobacco products or e-cigarettes) and one bystander cohabiting with the user
  Interventions: Other: No intervention
- Non-smokers and non-users (control): Smoke free households (participants should be adult (18 years old and above), non e-cigarette user (never or former e-cigarette user >1 month), non-user of any kind of tobacco product (never or former user >1 month), and other household members should not be users of tobacco products or e-cigarettes
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention; 1 week observational study

SUMMARY:
Objective: To investigate in real-life conditions passive exposure to aerosols from the use of e-cigarettes among people who cohabit with e-cigarette users. A secondary objective is to investigate passive exposure to emissions from the use of conventional cigarettes and heated tobacco products among people who cohabit with users of these tobacco products.

Study design: This is an observational study conducted in four types of households: a) Homes with one exclusive e-cigarette user and at least one non-user (non-smoker), and no other users of any type of tobacco products. In these homes, one non-user and one user will be included in the study as participants ("type A" homes); b) Homes with one exclusive heated tobacco product (HTP) user and at least one non-user (non-smoker), and no other users of any type of tobacco products or e-cigarettes. In these homes, one non-user and one user will be included in the study as participants ("type B" homes); c) Homes with one exclusive manufactured cigarette smoker (not roll-your-own) and at least one non-smoker, and no other users of any type of tobacco products or e-cigarettes. In these homes, one non-smoker and one smoker will be included in the study as participants ("type C" homes); and d) Homes where no one uses e-cigarettes or consumes any other type of tobacco products (smoke-free homes). In these homes, one adult volunteer will be included in the study as a participant ("type D" homes).

The study will be conducted in 4 countries: Greece (Athens), Italy (Milan), Spain (Barcelona) and the UK (Edinburgh). Overall, the sample in each participating country will consist of the types of participants mentioned above, with a total of 250 participants.

Measurements: Passive exposure to e-cigarette aerosols will be assessed by measuring particulate matter (PM2.5) and airborne nicotine in the main room of homes during 7 days. Participants' saliva samples will be collected for nicotine and cotinine assessment. In addition, participants will be asked to fill in a personal diary about the use of e-cigarettes, second-hand exposure to e-cigarette aerosols (SHA) and exposure to second-hand smoke (SHS) produced by the use of conventional cigarettes.

DETAILED DESCRIPTION:
Aims: The main objective of this study is to investigate in real-life conditions passive exposure to aerosols from the use of e-cigarettes among people who cohabit with e-cigarette users. A secondary objective is to investigate passive exposure to emissions from the use of conventional cigarettes and heated tobacco products among people who cohabit with users of these tobacco products.

Study design

This is an observational study conducted in four types of households:

1. Homes with one exclusive e-cigarette user and at least one non-user (non-smoker), and no other users of any type of tobacco products. In these homes, one non-user and one user will be included in the study as participants ("type A" homes).
2. Homes with one exclusive heated tobacco product (HTP) user and at least one non-user (non-smoker), and no other users of any type of tobacco products or e-cigarettes. In these homes, one non-user and one user will be included in the study as participants ("type B" homes).
3. Homes with one exclusive manufactured cigarette smoker (not roll-your-own) and at least one non-smoker, and no other users of any type of tobacco products or e-cigarettes. In these homes, one non-smoker and one smoker will be included in the study as participants ("type C" homes).
4. Homes where no one uses e-cigarettes or consumes any other type of tobacco products (smoke-free homes). In these homes, one adult volunteer will be included in the study as a participant ("type D" homes).

The study will be conducted in 4 countries: Greece (Athens), Italy (Milan), Spain (Barcelona) and the UK (Edinburgh).

Passive exposure to e-cigarette aerosols will be assessed by measuring particulate matter (PM2.5) and airborne nicotine in the main room of homes during 7 days. Participants' saliva samples will be collected for nicotine and cotinine assessment. In addition, participants will be asked to fill in a personal diary about the use of e-cigarettes, second-hand exposure to e-cigarette aerosols (SHA) and exposure to second-hand smoke (SHS) produced by the use of conventional cigarettes.

Fieldwork

Once in the participants' home:

1. After checking the inclusion and exclusion criteria, the participants will be re-informed (information was provided when contacting for the first time the participants) about the study (information sheet for participants) and will be asked to provide their informed written consent. They will be also informed about a reward for their participation after finishing the study (gift card to be used in a local cultural store with value of 15€).
2. Measurement of nicotine using active sampling will be initiated, lasting 30 min and record of smoking/use pattern if applicable using the home dossier.
3. The researcher will install the monitor with a filter for nicotine sampling that will be left at homes of the participants during the week of the study.
4. The researcher will administer to the participant the questionnaire about usual exposure to SHS and SHA (for all participants) and about consumption practices and habits (for users).
5. The participants will be instructed about the completion of the diary card that will be used to collect daily information about exposure to SHS and SHA (for all participants) and about patterns of smoking, e-cigarette or HTP use.
6. The first saliva sample will be collected under the supervision of the researcher.
7. AirVisual, an optical PM2.5 monitoring device, will be installed in the main room of the home. The participants will be instructed about its functioning and contact details for any questions will be provided in participant information leaflet.
8. The container for urine sample to be collected at the second visit after one week of the study with instructions on the procedures will be provided to the participants.
9. The participants will be informed that:

   * the researchers will be available for any queries during the study period and a contact phone number will be provided;
   * reminders to fill in the diary card will be sent via emails (SMS or the system chosen by the participant) every day; and
   * the researchers will make a follow-up telephone call during the study period
10. The researcher should inform about the day when the second visit should be done (after 7 days of the study) and confirm the time with the participants During the consequent 7 days

During 7 days of the study

The researcher will:

* call the participant to check the progress and resolve any queries, at the day 3 or 4 of the study.
* send a text message (SMS or other system) daily to remind to fill in the diary card
* send a text message in the morning of the day of the second visit to remind about urine sample collection

The participants will:

- fill in the diary card to record any exposure to SHA and/or SHS at home and other settings (for all participants) and e-cigarette, HTP use or smoking pattern (for e-cigarette, HTP users and smokers).

Second visit (7 days after first visit)

In the participants' homes, the researchers will:

* measure airborne nicotine with active sampling for 30 minutes (2nd measurement)
* review the diary cards with the participant(s) and collect them
* collect the AirVisual device and passive nicotine sampler
* collect a second saliva sample
* ask to the participant(s) for sample of e-liquid used (for e-cigarette users)
* collect the urine sample prepared by the participants (if applies)
* give the gift card to participants and ask them to sign the receipt form
* acknowledge the participation and remind that the feedback with the results of the study will be sent to them in approximately 6 months.

Data Management: All data from questionnaires, environmental measurements and saliva analysis will be managed by researchers from Tobacco Control Unit (UCT) of the Catalan Institute of Oncology.

Data will be collected in paper and will be digitalised in a protected database. All the samples (environmental, biological, and e-cigarette liquid) will have a unique code to be linked with the already anonymized data from the questionnaires, and this data will be stored in the same database. Only a selected number of pre-designated members of the research team (who will sign a confidentiality document) will have access to the database and the freezer. All data will be stored into a single database.

Selected personal data, including the names of respondents, will be collected separately to enable quality assurance procedures and to allow participants' willing to withdraw from participation in the study to have their records deleted from the database. This information will remain dissociated from the specific information generated in the experiments.

During the quality assurance procedures, Dr Esteve Fernández will obtain an anonymised copy of the database. The database will be held securely on a password protected file server at ICO. Dr Fernández will designate a limited number of researchers from UCT team or the consortium to access this database.

Access to personal data and withdrawal from the study: It will be made clear in the information (provided orally and in the information sheet) that the subjects are completely free to withdraw their records from participation in the study, regardless having had a gift compensation for their participation.

The consent given by participants in the project can be withdrawn at any time, without any explanation or justification. In this case, all data pertaining to the subjects will be destroyed, both in paper and digital supports.

At the end of the study, participants will receive the results from the environmental and biological measurements conducted as well as the overall results obtained for the entire study subjects. Summary data related to the entire project will be publicly disseminated once it has been processed and protected, without data that allow individual identification of participants. These summary results will be accessed through the project website or through publications related to this project.

Human cells/tissues: Biological samples (saliva and urine) will be collected after obtaining informed consent, in which it will be specified that these samples will be used only for the study aims, this is, the measurement of nicotine, cotinine and other metabolites of nicotine, metals and other markers of exposure to aerosols from e-cigarettes, but not for the use of the cells or genetic material also contained in the saliva. The remaining saliva and urine will be stored at the certified biobank (at ICO) and can be used for future determinations of compounds from cigarettes and e-cigarettes related with the objectives of this study.

Privacy and confidentiality: All personal information will be treated as confidential and will be stored in agreement with the current laws. The study will be conducted in accordance with the Good Clinical Practice Guidelines of the Declaration of Helsinki and the current legal regulation about confidentiality of data in the European Union (Regulation EU 2016/679 of the European Parliament and of the Council).

Environmental protection and safety: This study will require some exposure from the participants; however, this exposure will be the usual one and the participants will not be forced to any additional exposure given the observational nature of the study conducted. They will record the usual exposures without any intervention from the research team. Similarly, the researchers can be also exposed to emissions from tobacco products, but the total time of potential exposure is out of the range of potential health hazards produced by these exposures. All the researchers have been informed and have signed a written consent about their participation.

Incidental findings: In case that while reviewing the results from the chemical analysis of nicotine metabolites in saliva any unexpected abnormality is observed (what is called an "incidental finding"), the investigators will let the participant know. Depending on the type of incidental finding, the participant will be contacted by mail or by phone. The participant does not have an option to decline information about an incidental finding. The costs for any care that will be needed to diagnose or treat an incidental finding would not be paid for the research study. These costs would be the responsibility of the participant.

ELIGIBILITY:
Inclusion Criteria:

Non-e-cigarette and non-tobacco-product users

* Adult (18 years old and above)
* Non e-cigarette user (never or former e-cigarette user >1 month)
* Non-user of any kind of tobacco product (never or former user >1 month)
* [Only for type D homes]: other household members should not be users of tobacco products or e-cigarettes

E-cigarette users

* Adult (18 years old and above)
* E-cigarette exclusive user for at least 1 month
* Daily use of e-cigarettes inside home
* Cohabiting with at least one non-tobacco product nor e-cigarette user
* Other household members should not be users of any tobacco products or e-cigarettes

Heated tobacco product users

* Adult (18 years old and above)
* HTP exclusive user for at least 1 month
* Daily use of HTP inside home
* Cohabiting with at least one non-tobacco product nor e-cigarette user
* Other household members should not be users of tobacco products or e-cigarettes

Manufactured cigarette smoker

* Adult (18 years old and above)
* Manufactured cigarette exclusive smoker (not roll-your-own) for at least 6 months
* Daily smoking inside home
* Cohabiting with at least one non-tobacco product nor e-cigarette user
* Other household members should not be users of tobacco products or e-cigarettes

Exclusion Criteria:

For all participants:

• To be daily exposed to SHS from tobacco products or to SHA from e-cigarettes in places other than home.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Overall, the sample in each participating country will consist of these types of participants:
  Type A 20 e-cigarette users 20 non-users cohabiting with e-cigarette users Type B* 5 heated tobacco product users 5 non-users cohabiting with heated tobacco product users Type C 5 conventional cigarette smokers 5 non-smokers cohabiting with conventional cigarette smokers Type D 5 non-smokers/non-users living in smoke/e-cigarette free homes
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Airborne nicotine concentration (mg/m3) | 7 days
  Median airborne nicotine concentration (1h measurements with active sampling and 7-day continuous of passive sampling) in the home environment

SECONDARY OUTCOMES:
Particulate matter concentration (PM2.5; in mg/m3) | 7 days
  Median PM2.5 concentrations (7-day continuous) in the home environment
Nicotine, cotinine, TSNAs and propylene glycole concentrations in saliva samples (in ng/ml) | 1st day and the 7th day (pre-; post)
  Median concentrations of tobacco-related components in saliva samples
Metals, nicotine, cotinine and TSNAs concentrations in urine samples (in ng/ml) | One measurement; day 7 of the observational study
  Metals, nicotine, cotinine and TSNAs concentrations in urine samples (collected only in Spain and Italy)

CONTACTS AND LOCATIONS:
Overall Officials: Esteve Fernández, Dr, Principal Investigator — Catalan Institute of Oncology (ICO) // Bellvitge Biomedical Research Institute (IDIBELL)
Locations (1):
- Catalan Institute of Oncology, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: TackSHS Project at CORDIS — https://cordis.europa.eu/project/rcn/198790/factsheet/en